CLINICAL TRIAL: NCT01731379
Title: In Vivo Identification of Peripheral Nerve Bundles During Surgery Using Optical Spectroscopy Techniques - a Pilot Study
Brief Title: Optical Detection of Peripheral Nerve Bundles During Surgery
Acronym: NerveSpect
Status: Completed | Type: Observational
Sponsor: Philips Healthcare (Industry)
Collaborators: Philips Electronics Nederland B.V. acting through Philips CTO organization (Industry)
Responsible Party: Sponsor
Other Study IDs: NL 40893.031.12
Record Dates: First submitted 2012-11-16; First posted 2012-11-21 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Malignant Lymphoma of Lymph Nodes of Inguinal Region; Malignant Lymphoma of Lymph Nodes of Axillary; Malignant Lymphoma of Lymph Nodes of the Cervix; Carcinoma of Parotid Gland; Colon Rectal Cancer Tubulovillous Adenocarcinoma; Tumor of Soft Tissue of Head, Face and Neck
Keywords: spectroscopy; nerve; muscle; fat
MeSH Terms: conditions — Parotid Neoplasms; Facies; Platelet Glycoprotein IV Deficiency | interventions — Lymph Node Excision

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Surgical resections: Patients planned for elective inguinal, axillary or cervical lymph node dissection or parotidectomy, patients with rectal cancer undergoing rectal surgery and patients undergoing resection of a soft tissue tumour.
  Interventions: Procedure: Surgical resection

INTERVENTIONS:
Procedure: Surgical resection — Patients planned for elective inguinal, axillary or cervical lymph node dissection or parotidectomy , patients with rectal cancer undergoing rectal surgery and patients undergoing resection of a soft tissue tumour.
  Other Names: lymph node dissection; resection of parotid gland; rectal surgery; soft tumor resection

SUMMARY:
Investigation of application possibilities of optical spectroscopy within the field of surgical resection procedures to spare nerve tissue. Optical spectroscopy enables the possibility to specifically differentiate between different (human) tissues. The hypothesis is that incorporation of this technique into existing medical devices (e.g. medical blade) would enlarge the accuracy and reliability of these devices. Sparing of nerve bundles during surgery can lead to decreased postoperative morbidity rates.

DETAILED DESCRIPTION:
The aim of this pilot study is to prove that an investigational optical spectroscopy system can provide accurate identification of nerve tissue during surgery.

Primary Objective:

The goal of this pilot study is to evaluate whether optical spectroscopy is able to differentiate between nerve tissue and surrounding tissue.

Secondary Objective:

During the measurement procedure, possible improvements of the measurement hardware will be recorded and the handling of the optical spectroscopy system during surgery will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for elective inguinal, axillary or cervical lymph node dissection or parotidectomy , patients with rectal cancer undergoing rectal surgery and patients undergoing resection of a soft tissue tumour.
* Patients that have provided a signed informed consent
* Patients ≥ 18 years old

Exclusion Criteria:

• Patients with suspected sensitivity to light; e.g. patients who have had photodynamic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients are patients of the Netherlands Cancer Institute (NKI-AvL), who are scheduled for an elective inguinal, axillary or cervical lymph node dissection, or parotidectomy as well as patients with rectal cancer undergoing rectal surgery and patients undergoing resection of a soft tissue tumour.
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2012-12; Primary Completion 2014-01 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Differentiation between nerve tissue and its surrounding tissue | Day 0
  Statistical analysis of the difference between diffuse reflectance spectra obtained at nerve tissue and its surrounding tissue measurement locations

CONTACTS AND LOCATIONS:
Overall Officials: Theo Ruers, MD, Principal Investigator — Nederlands Kanker Instituut/Antonie van leeuwenhoek Ziekenhuis
Locations (1):
- Nederlands Kanker Instituut/Antonie van Leeuwenhoek Ziekenhuis, Amsterdam, North Holland, Netherlands